CLINICAL TRIAL: NCT06324448
Title: Self-administered Transcranial Direct Current Stimulation for Improving Single- and Dual-task Gait in Patients With Idiopathic Parkinson's Disease: A Prospective, Single-center, Double-blind, Exploratory, Randomized Controlled Trial
Brief Title: Self-administered tDCS for Improving Single- and Dual-task Gait in Patients With PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PD-tDCS-RCT
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; transcranial direct current stimulation; gait; dual-task
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary motor cortex (Experimental): The anodal electrode is positioned in the primary motor cortex (Cz) and the cathodal electrode on the right orbital frontal cortex (Fp2). The current increases to 2.0 mA over a period of 30 seconds, maintains 2.0 mA for 19 minutes, and decreases to 0 mA over 30 seconds.
  Interventions: Device: Transcranial direct current stimulation
- Left dorsolateral prefrontal cortex (Experimental): The anodal electrode is positioned in the left dorsolateral prefrontal cortex (F3) and the cathodal electrode on the right orbital frontal cortex (Fp2). The current increases to 2.0 mA over a period of 30 seconds, maintains 2.0 mA for 19 minutes, and decreases to 0 mA over 30 seconds.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS self-administered at home once a day for 28 consecutive days for a total of 28 sessions (one session consists of 20 minutes through two saline-soaked sponge electrodes (diameter 6cm) using the YMS-201B (Ybrain Inc, South Korea)).

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of self-administered transcranial direct current stimulation to improve the single- and dual-task gait in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a disease caused by dopamine deficiency in the striatum resulting from the loss of dopaminergic neuronal cells in the cerebral substantia. It is a progressive neurodegenerative disease characterized by motor symptoms including gait disturbance and balance instability. In the early stages of Parkinson's disease, dysfunction of the sensorimotor area of the basal ganglia typically occurs, leading to habitual control hurdles. Accordingly, cognitive efforts are required to perform habitual tasks such as walking, and the automaticity of walking is reduced. Dual-task performance involves a complex interplay of motor functions as well as cognitive functions such as attention and executive function. One way to potentially reduce the cost of dual-tasking and the negative effects of motor-cognitive interference is to consider improving the corresponding component, i.e., motor or cognitive function.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that can be used to change cortical activity. Recently, there has been growing attention on tDCS as an adjunct tool for rehabilitation. Several tDCS studies in patients with PD have reported the positive results of tDCS on motor and cognitive function. Most studies have examined changes before and after a single session of stimulation, with limited research verifying the cumulative and long-term effects of tDCS. Therefore, this study aims to investigate the efficacy and safety of self-administered transcranial direct current stimulation to improve the single- and dual-task gait in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as idiopathic Parkinson's disease by neurologists according to the UK Parkinson's Disease Society Brain Bank criteria
* modified Hoehn & Yahr stage 2, 2.5, or 3

Exclusion Criteria:

* History of seizure
* Metallic implants, such as cardiac pacemaker or an artificial cochlea
* Patients with inflammation, burns, or wounds in the stimulation area
* Parkinson's disease dementia; cut-off is < 7 of Korean-Montreal Cognitive Assessment for illiterate patients, < 13 for those educated for 0.5-3 years, < 16 for 4-6 years of education, < 19 for 7-9 years of education, and < 20 for 10 or more years of education.
* Severe dyskinesia or severe on-off phenomenon
* Plan to adjust medication at the time of screening
* Other neurological, orthopedic, or cardiovascular co-morbidities significantly affecting gait function
* Uncontrolled vestibular disease, orthopedic hypotension, or paroxysmal vertigo
* Pregnant or lactating patients
* Other comorbidities that make it difficult to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Timed-up and go test (sec) | Immediate post-intervention
Timed-up and go test under dual-task condition (sec) | Immediate post-intervention

SECONDARY OUTCOMES:
Dual-task effect (%) in Timed-up and go test | Immediate post-intervention
  Percentage of dual-task effect calculated by the difference between dual-task and single-task performance [Percentage of dual-task interference=(Dual-task performance - Single-task performance)/Single-task performance]
modified Attention Allocation Index (mAAI) in Timed-up and go test | Immediate post-intervention
  modified Attention Allocation Index (mAAI)=motor dual task effect(mDTE)-cognitive dual task effect (cogDTE)
Gait parameters | Immediate post-intervention
  Symmetric temporospatial parameters, Normal cadence, Decreased & intolerable walking velocity, Normal step length differential, Normal step length on both sides, Normal stride length on both sides, Normal swing phase & stance phase on both sides, Normal single support time & double support time on both sides, Slightly widened base of support on both sides, Increased foot angle on right side
Single-leg stance test | Immediate post-intervention
Stroop test | Immediate post-intervention
  The Stroop test evaluates attention, executive function, processing speed, and cognitive flexibility regarding an individual's ability to inhibit the habitual response.
Trail making test | Immediate post-intervention
  The trail-making test is a neuropsychological measure that assesses psychomotor speed, attention, sequencing, mental flexibility, and visual scanning.
New freezing of gait questionnaire (NFoGQ) | Immediate post-intervention
  NFoGQ consists of 6 items. Total score ranges from 0 to 24. the higher scores, the more negative results.
Geriatric depression scale (GDS)-short form | Immediate post-intervention
  The GDS Short Form contains 15 items. The higher the score, the more negative the result.
Timed-up and go test (sec) | Follow-up (1 month)
Timed-up and go test under dual-task condition (sec) | Follow-up (1 month)
Dual-task effect (%) in Timed-up and go test | Follow-up (1 month)
  Percentage of dual-task effect calculated by the difference between dual-task and single-task performance [Percentage of dual-task interference=(Dual-task performance - Single-task performance)/Single-task performance]
modified Attention Allocation Index (mAAI) in Timed-up and go test | Follow-up (1 month)
  modified Attention Allocation Index (mAAI)=motor dual task effect(mDTE)-cognitive dual task effect (cogDTE)
Gait parameters | Follow-up (1 month)
  Symmetric temporospatial parameters, Normal cadence, Decreased & intolerable walking velocity, Normal step length differential, Normal step length on both sides, Normal stride length on both sides, Normal swing phase & stance phase on both sides, Normal single support time & double support time on both sides, Slightly widened base of support on both sides, Increased foot angle on right side
Single-leg stance test | Follow-up (1 month)
Stroop test | Follow-up (1 month)
  The Stroop test evaluates attention, executive function, processing speed, and cognitive flexibility regarding an individual's ability to inhibit the habitual response.
Trail making test | Follow-up (1 month)
  The trail-making test is a neuropsychological measure that assesses psychomotor speed, attention, sequencing, mental flexibility, and visual scanning.
New freezing of gait questionnaire (NFoGQ) | Follow-up (1 month)
  NFoGQ consists of 6 items. Total score ranges from 0 to 24. the higher scores, the more negative results.
Geriatric depression scale (GDS)-short form | Follow-up (1 month)
  The GDS Short Form contains 15 items. The higher the score, the more negative the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea